CLINICAL TRIAL: NCT07405619
Title: Quality Assessment of Anterior Composite Restorations: Clinical Examination Versus Three Digital Photographic Techniques
Brief Title: Quality Assessment of Anterior Composite Restorations
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Yildiz Telatar, Recep Tayyip Erdoğan University-RIZE, Recep Tayyip Erdogan University
Other Study IDs: 2023/137
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Composite Resins
Keywords: anterior composite restorations; digital photography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Smartphone Photography — This study evaluates the diagnostic performance of three different digital imaging protocols compared to a physical clinical examination.

SUMMARY:
Evaluation of Intraoral Smartphone Photography for Anterior Restorations Purpose The goal of this observational study was to determine if intraoral digital photography-captured using modern smartphones-can accurately assess the quality of dental fillings (anterior composite restorations) compared to traditional in-person clinical exams.

DETAILED DESCRIPTION:
Evaluating the longevity and quality of dental restorations is a cornerstone of restorative dentistry. Traditionally, the World Dental Federation (FDI) criteria are applied during a physical clinical examination. However, the rise of teledentistry and the accessibility of high-resolution mobile imaging have created a need to validate digital photography as a diagnostic tool. This study investigates whether the convenience of smartphone photography can match the diagnostic "gold standard" of a clinical chairside exam and the technical "gold standard" of a professional DSLR camera.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Primary teeth, unrestored teeth, and teeth with amalgam, glass ionomer, or indirect restorations

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included 185 anterior teeth with composite restorations from individuals aged 18-64
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
Diagnostic Agreement for FDI Final Scores | At the time of the single clinical assessment (cross-sectional).
  The level of agreement between each digital photography method and the clinical examination (Gold Standard) for the overall restoration status. Restorations are categorized into three final scores: Intact, Requires Repair, or Needs Replacement based on World Dental Federation (FDI) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP

REFERENCES:
- [Result] Opdam NJM, Collares K, Hickel R, Bayne SC, Loomans BA, Cenci MS, Lynch CD, Correa MB, Demarco F, Schwendicke F, Wilson NHF. Clinical studies in restorative dentistry: New directions and new demands. Dent Mater. 2018 Jan;34(1):1-12. doi: 10.1016/j.dental.2017.08.187. Epub 2017 Sep 20. PMID 28941587